CLINICAL TRIAL: NCT02331004
Title: Effectiveness of an Intervention Program for Fine Motor Skills in Institutionalized Elderly Residents: a Randomized Clinical Trial
Brief Title: Effectiveness of an Intervention Program for Fine Motor Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Encarnación Aguilar Ferrandiz, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fine motor skills
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hand Injuries
Keywords: Frail Elderly; Motor Skills; Upper Extremity
MeSH Terms: conditions — Hand Injuries | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention for fine motor skills (Active Comparator): Implementation of an well known activity to improve the function of upper extremities
  Interventions: Other: Intervention for fine motor skills
- Support to activities of daily living (Placebo Comparator): Performing of general activities planned in the centres where the participants are included
  Interventions: Other: Support to activities of daily living

INTERVENTIONS:
Other: Intervention for fine motor skills — Implementation of an well known activity to improve the function of upper extremities
  Other Names: Performing of a specific manual activity
  Arms: Intervention for fine motor skills
Other: Support to activities of daily living — Participants are supported and orientated when they are performing some activity of daily living scheduled by the institution
  Other Names: Performing of activities of daily living
  Arms: Support to activities of daily living

SUMMARY:
Investigators have created a protocol of intervention to treating the general disability of upper limbs.

DETAILED DESCRIPTION:
A protocol of intervention for fine motor skills will be performed on institutionalized elderly people.

This protocol consist on implementation of a manual activity that it is well known in the clinical setting.

This activity will enhance several skills such as strength, coordination of upper limbs, range of motion, general auto-efficacy and the quality of life.

The intervention or rehabilitation will be implemented for two month.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized elderly people, on a full or part-time.
* Voluntary participation.

Exclusion Criteria:

* Cognitive impairment (< 23 in normal school population and < 20 points with a low education or illiteracy, in Spanish validation of Mini-Mental State Examination (MMSE)).
* Postural control problems.
* Balance disorders, while the subject is seated.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Disability of the Arm, Shoulder and Hand (DASH) questionnaire at 8 weeks | Eight weeks
Change from Baseline in Disability of the Arm, Shoulder and Hand (DASH) questionnaire at 16 weeks | Sixteen weeks

SECONDARY OUTCOMES:
Change from Baseline in General self-efficacy at 8 weeks | Eight weeks
Change from Baseline in General self-efficacy at 16 weeks | Sixteen weeks
Change from Baseline in Purdue Pegboard Tests at 8 weeks | Eight weeks
Change from Baseline in Purdue Pegboard Tests at 16 weeks | Sixteen weeks
Change from Baseline in finger goniometer at 8 weeks | Eight weeks
  Active and passive measures of motion in first, second and fifth fingers of dominant hand will be recorded .
Change from Baseline in finger goniometer at 16 weeks | Sixteen weeks
  Active and passive measures of motion in first, second and fifth fingers of dominant hand will be recorded .
Change from Baseline in Pinch Gauge at 8 weeks | Eight weeks
Change from Baseline in Pinch Gauge at 16 weeks | Sixteen weeks
Change from Baseline in Short-Form health survey questionnaire (SF-36) at 8 weeks | Eight weeks
Change from Baseline in Short-Form health survey questionnaire (SF-36) at 16 weeks | Sixteen weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mª Encarnacion ME Aguilar, PdH, Principal Investigator — Universidad de Granada
Locations (1):
- Maria Encarnación Aguilar Ferrandiz, Granada, Granada, Spain